CLINICAL TRIAL: NCT04798976
Title: Personalized Evidence-based Treatment Improves Survival in Patients With Invasive Breast Cancer
Brief Title: Personalized Evidence-based Treatment in Patients With Invasive Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Center of Personalized Medicine, Pirogova (Other)
Collaborators: Center for New Medical Technologies, Novosibirsk, Russia (Other); I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Evgeny Pokushalov, Director for research and development, Center of Personalized Medicine, Pirogova
Other Study IDs: 20210312
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer-specific Survival
MeSH Terms: interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CDSS (MedicBK) Analysis
  Interventions: Drug: neoadjuvant/adjuvant therapy
- Core Laboratory Analysis
  Interventions: Drug: neoadjuvant/adjuvant therapy

INTERVENTIONS:
Drug: neoadjuvant/adjuvant therapy — chemotherapy/endocrine therapy/surgery/radiotherapy

SUMMARY:
A population-based case-cohort study of breast cancer-specific survival among all first invasive breast cancer cases

ELIGIBILITY:
Inclusion Criteria:

All women with stage I-III disease who survived at least 12 months post-diagnosis

Exclusion Criteria:

Unknown cause of death Treatment outside the region (thus precluding the treatment assessment)

Max Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All first invasive breast cancer cases from a National Cancer Registry
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
The percentage of guideline-consistent and personalized EBM recommendations | 3-year
  The percentage of guideline-consistent and personalized EBM recommendations acted on by clinicians in patients with first invasive breast cancer. All discrepancies between routine and CDSS-recommended treatment resulting in frame of guideline-consistent therapy and personalized EBM therapy will be adjudicated by core laboratory.

SECONDARY OUTCOMES:
Breast cancer-specific survival | 3-year
  All deaths due to breast cancer-related causes
Quantify the performance of the CDSS (MedicBK) algorithm | 3-year
  Quantify the performance of the CDSS (MedicBK) algorithm for presents treatment suggestions in frame of guideline-based therapy and personalized EBM therapy: the sensitivity, specificity, NPV, and PPV
Predictors | 3-year
  Predictors of guideline-consistent and personalized EBM adherence

CONTACTS AND LOCATIONS:
Locations (1):
- Evgeny Pokushalov, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: Undecided